CLINICAL TRIAL: NCT00666536
Title: A Multicenter, Randomized, Double Blind, Parallel Design Trial to Evaluate the Blood Pressure Lowering Efficacy Comparing Moderate Versus Aggressive Treatment Regimen of Valsartan + Amlodipine in Patients Uncontrolled on ARB Monotherapy
Brief Title: The Effects of Moderate vs. Aggressive Treatment With Valsartan + Amlodipine on Patients With Hypertension Uncontrolled by Angiotensin-Receptor Blocker (Herein, ARB) Monotherapy
Acronym: EXTRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAA489AUS02
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Results first posted 2010-12-10 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
Keywords: Hypertension; adults; Valsartan + Amlodipine; Angiotensin Receptor Blockers
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aggressive treatment regimen (5/320 mg to 10/320 mg) (Active Comparator): Valsartan + Amlodipine, daily: 320 mg + 5 mg (2 weeks); Valsartan + Amlodipine, daily: 320 mg + 10 mg (2 weeks); Valsartan + Amlodipine and Hydrochlorothiazide, daily: 320 mg + 10 mg and 12.5 mg (4 weeks); Valsartan + Amlodipine and Hydrochlorothiazide, daily: 320 mg + 10 mg and 12.5 mg or 25 mg (optional titration) (4 weeks)
  Interventions: Drug: valsartan and amlodipine
- Moderate treatment regimen (5/160 mg) (Active Comparator): Valsartan + Amlodipine, daily dose: 160 mg + 5 mg (4 weeks); Valsartan + Amlodipine and Hydrochlorothiazide, daily: 160 mg + 5 mg and 12.5 mg (4 weeks); Valsartan + Amlodipine and Hydrochlorothiazide, daily: 160 mg + 5 mg and 12.5 mg or 25 mg (optional titration) (4 weeks)
  Interventions: Drug: valsartan and amlodipine

INTERVENTIONS:
Drug: valsartan and amlodipine
  Arms: Aggressive treatment regimen (5/320 mg to 10/320 mg)
Drug: valsartan and amlodipine
  Arms: Moderate treatment regimen (5/160 mg)

SUMMARY:
The purpose of this trial is to compare blood pressure lowering efficacy of moderate Valsartan + Amlodipine treatment regimen (160 / 5 mg) with that of aggressive regimen (320 / 10 mg) in patients uncontrolled on ARB monotherapy, other than Valsartan

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients
* 18 Years of age or older
* Mean Sitting Systolic Blood Pressure (the top number) greater than or equal to 150 mmHg and lower than 200 mmHg while on Angiotensin-Receptor Blocker monotherapy for a minimum period of 28 days prior to randomization

Exclusion Criteria:

* Mean Sitting Systolic Blood Pressure (the top number) greater than or equal to 200 mmHg and/or Mean Sitting Diastolic Blood Pressure greater than or equal to 120 mmHg
* Transient ischemic attack (mini-stroke), myocardial infarction (heart attack), all types of revascularization procedures in the last 6 months
* Treatment with valsartan or any combination antihypertensive treatment with 28 days prior to screening (Visit 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Oparil, MD et al, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Egan Healthcare, Metairie, Louisiana, United States

REFERENCES:
- [Result] Oparil S, Giles T, Ofili EO, Pitt B, Seifu Y, Hilkert R, Samuel R, Sowers JR. Moderate versus intensive treatment of hypertension with amlodipine/valsartan for patients uncontrolled on angiotensin receptor blocker monotherapy. J Hypertens. 2011 Jan;29(1):161-70. doi: 10.1097/HJH.0b013e32834000a7. PMID 21045734
- [Derived] Giles TD, Oparil S, Ofili EO, Pitt B, Purkayastha D, Hilkert R, Samuel R, Sowers JR. The role of ambulatory blood pressure monitoring compared with clinic and home blood pressure measures in evaluating moderate versus intensive treatment of hypertension with amlodipine/valsartan for patients uncontrolled on angiotensin receptor blocker monotherapy. Blood Press Monit. 2011 Apr;16(2):87-95. doi: 10.1097/MBP.0b013e328344c713. PMID 21386706

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 369 and 359 are the total randomized patients by treatment groups respectively. In the baseline measures tables 366 and 357 are the total patients for the ITT population by treatment group.
Period: Overall Study
Arm/Group | Aggressive Treatment Regimen (5/320 mg to 10/320 mg) | Moderate Treatment Regimen (5/160 mg)
Started | 369 | 359
Completed | 336 | 322
Not Completed | 33 | 37
Not completed — Adverse Event | 9 | 19
Not completed — Unsatisfactory therapeutic effect | 2 | 0
Not completed — Protocol deviation(s) | 8 | 6
Not completed — Withdrawal by Subject | 10 | 9
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aggressive Treatment Regimen (5/320 mg to 10/320 mg) | Moderate Treatment Regimen (5/160 mg) | Total
Number analyzed (Participants) | 366 | 357 | 723
Age, Customized [Number; unit: participants]
  < 65 years | 302 | 292 | 594
  >=65 years | 64 | 65 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (10.98) | 55.0 (10.98) | 54.7 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 157 | 314
  Male | 209 | 200 | 409

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in Mean Sitting Systolic Blood Pressure (MSSBP)
Time Frame: Baseline and Week 4
Population: Intent to treat (ITT), Last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aggressive Treatment Regimen (5/320 mg to 10/320 mg) | Moderate Treatment Regimen (5/160 mg)
Number analyzed (Participants) | 366 | 357
mmHg
  Baseline MSSBP | 163.9 (11.85) | 163.3 (11.40)
  Week 4 MSSBP | 140.9 (14.61) | 144.4 (14.21)
  Change From Baseline to Week 4 in MSSBP | -23.0 (14.60) | -18.9 (13.92)

2. Secondary Outcome: Percentage of Patients Achieving the Blood Pressure (BP) Goal of < 140/90 mmHg at Weeks 2,4,8 and 12
Time Frame: Weeks 2, 4, 8 and 12
Population: Intent to treat (ITT), Last observation carried forward (LOCF)
Measure: Number; unit: Percentage of Patients
Arm/Group | Aggressive Treatment Regimen (5/320 mg to 10/320 mg) | Moderate Treatment Regimen (5/160 mg)
Number analyzed (Participants) | 366 | 357
Percentage of Patients
  Week 2 | 25.1 | 25.8
  Week 4 | 43.7 | 31.1
  Week 8 | 61.7 | 46.2
  Week 12 | 59.8 | 50.7

3. Secondary Outcome: Change From Baseline to Week 4 in Mean Sitting Diastolic Blood Pressure (MSDBP)
Time Frame: Baseline and Week 4
Population: Intent to treat (ITT), Last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aggressive Treatment Regimen (5/320 mg to 10/320 mg) | Moderate Treatment Regimen (5/160 mg)
Number analyzed (Participants) | 366 | 357
mmHg
  Baseline MSDBP | 95.5 (11.19) | 95.0 (10.33)
  Week 4 MSDBP | 84.8 (11.47) | 86.2 (9.6)
  Change From Baseline to Week 4 in MSDBP | -10.7 (9.39) | -8.8 (9.08)

4. Secondary Outcome: Change From Baseline to Weeks 2, 8 and 12 in MSSBP
Time Frame: Baseline and Weeks 2, 8 and 12
Population: Intent to treat (ITT), Last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aggressive Treatment Regimen (5/320 mg to 10/320 mg) | Moderate Treatment Regimen (5/160 mg)
Number analyzed (Participants) | 366 | 357
mmHg
  Baseline MSSBP | 163.9 (11.85) | 163.3 (11.40)
  Week 2 MSSBP | 147.0 (14.93) | 146.0 (14.80)
  Change From Baseline to Week 2 in MSSBP | -16.9 (13.94) | -17.3 (13.80)
  Week 8 MSSBP | 136.0 (15.27) | 140.5 (15.91)
  Change From Baseline to Week 8 in MSSBP | -27.9 (16.08) | -22.8 (16.15)
  Week 12 MSSBP | 135.7 (14.97) | 139.2 (15.63)
  Change From Baseline to Week 12 in MSSBP | -28.1 (16.59) | -24.1 (16.07)

5. Secondary Outcome: Change From Baseline to Weeks 2, 8 and 12 in MSDBP
Time Frame: Baseline and Weeks 2, 8 and 12
Population: Intent to treat (ITT), Last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aggressive Treatment Regimen (5/320 mg to 10/320 mg) | Moderate Treatment Regimen (5/160 mg)
Number analyzed (Participants) | 366 | 357
mmHg
  Baseline MSDBP | 95.5 (11.19) | 95.0 (10.33)
  Week 2 MSDBP | 88.2 (10.93) | 87.1 (10.38)
  Change From Baseline to Week 2 in MSDBP | -7.3 (8.51) | -7.9 (9.66)
  Week 8 MSDBP | 81.6 (11.15) | 84.0 (11.39)
  Change From Baseline to Week 8 in MSDBP | -13.9 (9.97) | -11.0 (10.33)
  Week 12 MSDBP | 81.5 (10.62) | 83.8 (10.61)
  Change From Baseline to Week 12 in MSDBP | -14.0 (10.41) | -11.2 (10.48)

6. Secondary Outcome: Percentage of Patients Achieving BP Goal of MSSBP < 140mmHg at Weeks 2, 4, 8 and 12
Time Frame: Weeks 2, 4, 8 and 12
Population: Intent to treat (ITT), Last observation carried forward (LOCF)
Measure: Number; unit: Percentage of Patients
Arm/Group | Aggressive Treatment Regimen (5/320 mg to 10/320 mg) | Moderate Treatment Regimen (5/160 mg)
Number analyzed (Participants) | 366 | 357
Percentage of Patients
  Week 2 | 31.1 | 32.5
  Week 4 | 49.2 | 37.5
  Week 8 | 66.1 | 49.6
  Week 12 | 62.8 | 55.7

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Aggressive Treatment Regimen (5/320 mg to 10/320 mg) | Moderate Treatment Regimen (5/160 mg)
Serious Adverse Events (participants affected / at risk) | 4/369 | 10/359
Other Adverse Events (participants affected / at risk) | 50/369 | 29/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aggressive Treatment Regimen (5/320 mg to 10/320 mg) (N=369) | Moderate Treatment Regimen (5/160 mg) (N=359)
Angina pectoris (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Palpitations (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aggressive Treatment Regimen (5/320 mg to 10/320 mg) (N=369) | Moderate Treatment Regimen (5/160 mg) (N=359)
Oedema peripheral (General disorders) | 32 | 16
Dizziness (Nervous system disorders) | 19 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.